CLINICAL TRIAL: NCT02481310
Title: A Phase I-II Trial of DA-EPOCH-R Plus Ixazomib as Frontline Therapy for Patients With MYC-aberrant Lymphoid Malignancies: The DACIPHOR Regimen
Brief Title: Combination Chemotherapy, Rituximab, and Ixazomib Citrate in Treating Patients With Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 14H09; NCI-2015-00400 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16042; STU00200596; NU 14H09 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-06-25 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Adult Burkitt Lymphoma; B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Burkitt Lymphoma; Diffuse Large B-Cell Lymphoma; MYC Gene Mutation; Plasmablastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Plasmablastic Lymphoma | interventions — Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; ixazomib; Methotrexate; merphos; Prednisone; deltacortene; prednylidene; Rituximab; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy, rituximab, ixazomib) (Experimental): INDUCTION:
  Patients receive ixazomib citrate PO on day 1 and day 8 or 15; etoposide IV, vincristine sulfate IV, and doxorubicin hydrochloride IV continuously over 96 hours on days 1-4; prednisone PO BID on days 1-5; rituximab IV should be started at 50 mg/hr, and increased in 50-mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr on day 1; and cyclophosphamide IV over 90 minutes on day 5.
  CNS PROPHYLAXIS:
  Patients with a negative LP receive methotrexate IT once per course. Patients with a positive LP receive methotrexate IT or intraventricularly OR cytarabine IT or intraventricularly OR methotrexate IT or intraventricularly, cytarabine IT or intraventricularly, and therapeutic hydrocortisone IT or intraventricularly.
  MAINTENANCE:
  Patients not treated with consolidative SCT, receive ixazomib citrate PO BID on days 1, 8, and 15. Treatment repeats every 28 days for up to one year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Drug: Prednisone; Biological: Rituximab; Drug: Therapeutic Hydrocortisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT or intraventricularly
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IT or intraventricularly
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Drug: Therapeutic Hydrocortisone — Given IT or intraventricularly
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; HYDROCORTISONE; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
The purpose of this study is to evaluate the effects, good and bad of a new drug called ixazomib (also called MLN9708), when it is given along with a common treatment combination, called Dose-Adjusted EPOCH-R (DA-EPOCH-R, for short). This is a type of study called a phase I/II trial. In the phase I part, the dose of the study drug (ixazomib) will be adjusted (either up or down) to find the maximum (highest) dose that does not cause excessive (too many) harmful side effects. In the phase II part, this dose of ixazomib will be given at the maximum safe dose found in phase I. In both phase I and II, DA-EPOCH-R will be adjusted between cycles depending on how blood cell levels are affected between cycles. Ixazomib is considered investigational because it is not approved by the U.S. Food and Drug Administration (FDA). DA-EPOCH-R is a combination chemotherapy treatment developed over the last 14-15 years, and each of the drugs in this regimen is FDA-approved and considered part of the standard of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of ixazomib (ixazomib citrate) given with dose-adjusted etoposide, prednisone, vincristine (vincristine sulfate), cyclophosphamide, doxorubicin (doxorubicin hydrochloride), and rituximab (DA-EPOCH-R) in patients with aggressive, v-myc avian myelocytomatosis viral oncogene homolog (MYC)-aberrant lymphoid malignancies, and to determine the recommended phase II dose (RP2D) of the combination. (Phase I) II. To evaluate the efficacy, as measured by 12-month progression free survival (PFS), of ixazomib given with DA-EPOCH-R in patients with aggressive, MYC-aberrant lymphoid malignancies. (Phase II)

SECONDARY OBJECTIVES:

I. Further evaluate the frequency and severity of toxicity. II. Further evaluate the clinical efficacy, as measured by response rate and overall survival (OS).

III. Assess the predictive value of fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) scans on PFS.

TERTIARY OBJECTIVES:

I. Determine the impact of cell of origin (COO) upon response rate, PFS, and OS.

II. Assess the feasibility and outcomes of consolidation stem cell transplant (SCT).

OUTLINE: This is a phase I, dose-escalation study of ixazomib citrate followed by a phase II study.

INDUCTION:

Patients receive ixazomib citrate orally (PO) on day 1 and day 8 or 15; etoposide intravenously (IV), vincristine sulfate IV, and doxorubicin hydrochloride IV continuously over 96 hours on days 1-4; prednisone PO twice daily (BID) on days 1-5; rituximab IV should be started at 50 mg/hr, and increased in 50-mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr on day 1; and cyclophosphamide IV over 90 minutes on day 5.

CENTRAL NERVOUS SYSTEM (CNS) PROPHYLAXIS:

Patients with a negative lumbar puncture (LP) receive methotrexate intrathecally (IT) once per course. Patients with a positive LP receive methotrexate IT or intraventricularly OR cytarabine IT or intraventricularly OR methotrexate IT or intraventricularly, cytarabine IT or intraventricularly, and therapeutic hydrocortisone IT or intraventricularly.

MAINTENANCE:

Patients not treated with consolidative SCT, receive ixazomib citrate PO BID on days 1, 8, and 15. Treatment repeats every 28 days for up to one year (or as long as deriving benefit) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological diagnosis of any of the following (all stages allowed):

  * Diffuse large b-cell lymphoma (DLBCL) (including transformation from a previously indolent non-Hodgkin lymphoma [NHL], so long as no prior systemic treatment was given for the indolent NHL)
  * B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma
  * Burkitt lymphoma
  * MYC+ plasmablastic lymphoma by histology
* Patients must have measurable disease (defined as >= 1.5 cm in diameter)
* Patients must have MYC-rearrangement, as determined by fluorescent in-situ hybridization (FISH) (does not require central review)
* The following results must be available or pending at time of registration, though results will not affect enrollment/treatment:

  * B-cell chronic lymphocytic leukemia (CLL)/lymphoma (BCL)-2 rearrangement by FISH
  * BCL-6 rearrangement by FISH NOTE: although not required, it is encouraged that MYC and BCL-2 be measured by immunohistochemistry (IHC) and clearly documented
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelets >= 75,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN); NOTE: exceptions can be granted from principal investigator (PI) for instances of Gilbert's disease, and/or primarily indirect bilirubinemia, if due to recent transfusion and/or hemolysis
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SPGT]) =< 3 X institutional ULN
* Calculated creatinine clearance >= 30 mL/min
* NOTE: platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before registration; these requirements do not apply to those with marrow involvement of lymphoma (any extent)
* Female patients must meet one of the following criteria:

  * Postmenopausal for at least 1 year prior to registration
  * Surgically sterile
  * Of childbearing potential and agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug
  * Of childbearing potential and agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject NOTE: periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject NOTE: periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Females of child-bearing potential (FOCBP) must have a negative pregnancy test within # days prior to registration on study
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had more than one cycle of prior chemoimmunotherapy for diagnosis of NHL are not eligible; NOTE: such patients must have fully recovered (ie, =< grade 1 toxicity) from the reversible effects of prior chemotherapy before starting treatment on the current protocol
* Patients who have had major surgery within 4 weeks prior to registration are not eligible
* Patients who have had radiotherapy within 14 days before registration are not eligible; NOTE: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Patients who have an infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment are not eligible
* Patients who have evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months are not eligible
* Patients who have undergone systemic treatment, within 14 days prior to registration, with strong inhibitors of cytochrome P450 superfamily (CYP)1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort are not eligible
* Patients who have a clinically active hepatitis B or C virus infection are not eligible; NOTE: those with evidence of exposure to hepatitis B virus (HBV) may enroll so long as HBV viral load is negative AND subject is willing/able to take appropriate antiviral prophylaxis to prevent reactivation
* Patients with any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol are not eligible
* Patients who have a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent are not eligible
* Patients who have a known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing are not eligible
* Patients who have been diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease are not eligible; NOTE: Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patients who have >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period are not eligible
* Patients who are participating in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of registration and throughout the duration of this trial are not eligible
* Female patients who are nursing or have a positive pregnancy test during screening are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2024-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pro, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Tufts University, Medford, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Karmali R, Galvez C, Hamadani M, Gordon L, Winter J, Ma S, Nelson V, Fenske TS, Shah NN, Jagadeesh D, Klein A, Helenowski I, Chen R, Mi X, Petrich A, Evens AM, Pro B. A phase 1-2 trial of DA-EPOCH-R plus ixazomib for MYC-aberrant lymphoid malignancies: the DACIPHOR regimen. Blood Adv. 2024 Apr 9;8(7):1612-1620. doi: 10.1182/bloodadvances.2023011369. PMID 38237077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on Aug 24, 2015 with the first patient being enrolled and starting treatment on 10.28.2015. The study closed to any further accrual on October 1sts 2019 with 38 patients enrolled on study. The study closed prior to reaching full accrual goal of up to 55 patients.
Pre-assignment Details: First patient was enrolled to Cohort 1. Second patient enrolled to Cohort 2. Third patient enrolled to Cohort 3. Forth and fifth patient enrolled to Cohort 2. All further patients enrolled to phase II (same dose as Cohort 2).
Groups:
- Treatment- Cohort 1(Combination Chemotherapy, Rituximab, Ixazomib 2.3 mg): INDUCTION:
  Patients receive ixazomib citrate PO on day 1 and day 8 or 15; etoposide IV, vincristine sulfate IV, and doxorubicin hydrochloride IV continuously over 96 hours on days 1-4; prednisone PO BID on days 1-5; rituximab IV should be started at 50 mg/hr, and increased in 50-mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr on day 1; and cyclophosphamide IV over 90 minutes on day 5.
  CNS PROPHYLAXIS:
  Patients with a negative LP receive methotrexate IT once per course. Patients with a positive LP receive methotrexate IT or intraventricularly OR cytarabine IT or intraventricularly OR methotrexate IT or intraventricularly, cytarabine IT or intraventricularly, and therapeutic hydrocortisone IT or intraventricularly.
  MAINTENANCE:
  Patients not treated with consolidative SCT, receive ixazomib citrate PO BID on days 1, 8, and 15. Treatment repeats every 28 days for up to one year in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Cytarabine: Given IT or intraventricularly
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ixazomib Citrate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IT or intraventricularly
  Prednisone: Given PO
  Rituximab: Given IV
  Therapeutic Hydrocortisone: Given IT or intraventricularly
  Vincristine Sulfate: Given IV
- Treatment Cohort 2 and Phase II (Combination Chemotherapy, Rituximab, Ixazomib 3 mg); Treatment - Cohort 3 (Combination Chemotherapy, Rituximab, Ixazomib 4 mg): NDUCTION:
  Patients receive ixazomib citrate PO on day 1 and day 8 or 15; etoposide IV, vincristine sulfate IV, and doxorubicin hydrochloride IV continuously over 96 hours on days 1-4; prednisone PO BID on days 1-5; rituximab IV should be started at 50 mg/hr, and increased in 50-mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr on day 1; and cyclophosphamide IV over 90 minutes on day 5.
  CNS PROPHYLAXIS:
  Patients with a negative LP receive methotrexate IT once per course. Patients with a positive LP receive methotrexate IT or intraventricularly OR cytarabine IT or intraventricularly OR methotrexate IT or intraventricularly, cytarabine IT or intraventricularly, and therapeutic hydrocortisone IT or intraventricularly.
  MAINTENANCE:
  Patients not treated with consolidative SCT, receive ixazomib citrate PO BID on days 1, 8, and 15. Treatment repeats every 28 days for up to one year in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Cytarabine: Given IT or intraventricularly
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ixazomib Citrate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IT or intraventricularly
  Prednisone: Given PO
  Rituximab: Given IV
  Therapeutic Hydrocortisone: Given IT or intraventricularly
  Vincristine Sulfate: Given IV
Period: Induction Treatment (6 Cycles)
Arm/Group | Treatment- Cohort 1(Combination Chemotherapy, Rituximab, Ixazomib 2.3 mg) | Treatment Cohort 2 and Phase II (Combination Chemotherapy, Rituximab, Ixazomib 3 mg) | Treatment - Cohort 3 (Combination Chemotherapy, Rituximab, Ixazomib 4 mg)
Started | 1 | 36 | 1
Reached First Evaluable Response | 1 | 34 | 1
Complete 6 Cycles | 1 | 30 | 1
Completed | 1 | 30 | 1
Not Completed | 0 | 6 | 0
Period: Maintenance Treatment
Arm/Group | Treatment- Cohort 1(Combination Chemotherapy, Rituximab, Ixazomib 2.3 mg) | Treatment Cohort 2 and Phase II (Combination Chemotherapy, Rituximab, Ixazomib 3 mg) | Treatment - Cohort 3 (Combination Chemotherapy, Rituximab, Ixazomib 4 mg)
Started (Maintenance treatment can continue for up to one year or longer for continued clinical benefit if approved.) | 1 | 21 (9 patients that competed induction did not start maintenance treatment.) | 1
Started Maintenance Treatment | 1 | 21 | 1
Completed | 1 | 21 | 1
Not Completed | 0 | 0 | 0
Period: Follow up
Arm/Group | Treatment- Cohort 1(Combination Chemotherapy, Rituximab, Ixazomib 2.3 mg) | Treatment Cohort 2 and Phase II (Combination Chemotherapy, Rituximab, Ixazomib 3 mg) | Treatment - Cohort 3 (Combination Chemotherapy, Rituximab, Ixazomib 4 mg)
Started (All patients that are treated with at least one dose of study drug go into the follow up period.) | 1 | 32 (2 patients died prior to entering follow up, 1 patient withdrew consent and 1 patient currently on treatment.) | 1
Completed | 1 | 29 | 1
Not Completed | 0 | 3 | 0
Not completed — Still in follow up | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment- Cohort 1(Combination Chemotherapy, Rituximab, Ixazomib 2.3 mg) | Treatment Cohort 2 and Phase II (Combination Chemotherapy, Rituximab, Ixazomib 3 mg) | Treatment - Cohort 3 (Combination Chemotherapy, Rituximab, Ixazomib 4 mg) | Total
Number analyzed (Participants) | 1 | 36 | 1 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 25 | 0 | 25
  >=65 years | 1 | 11 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 11 | 0 | 11
  Male | 1 | 25 | 1 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 35 | 1 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3
  White | 1 | 33 | 1 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Recommended Phase II Dose (RP2D) of Ixazomib in Combination With DA-EPOCH-R.
Description: The RP2D will be determined by the evaluation of dose-limiting toxicities (DLT) to find the Maximum Tolerated Dose (MTD) which will constitute the RP2D. DLTs will be defined as the occurrence of ≥ Grade 3 toxicity experienced during the first cycle (3 weeks or 21 days) of study treatment, will be determined, except for cytopenias.
  The dose of ixazomib will start at 2.3 mg weekly (for phase I patients) when given concurrently with DA-EPOCH-R. Single-subject cohorts (escalating in ixazomib dose) will be enrolled until the MTD is encountered, after which expansion to 3-subject cohorts will be undertaken. The MTD from phase I will equate the RP2D for ixazomib given in conjunction with DA-EPOCH-R.
Time Frame: The first 21 days of treatment
Population: 1 patient enrolled at 2.3 mg of ixazomib, 3 patients enrolled at 3 mg of ixazomib, 1 patient enrolled at 4 mg ixazomib in phase I were evaluable for this endpoint.
Measure: Number; unit: mg
Groups:
- Treatment (Combination Chemotherapy, Rituximab, Ixazomib): INDUCTION:
  Patients receive ixazomib citrate PO on day 1 and day 8 or 15; etoposide IV, vincristine sulfate IV, and doxorubicin hydrochloride IV continuously over 96 hours on days 1-4; prednisone PO BID on days 1-5; rituximab IV should be started at 50 mg/hr, and increased in 50-mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr on day 1; and cyclophosphamide IV over 90 minutes on day 5.
  CNS PROPHYLAXIS:
  Patients with a negative LP receive methotrexate IT once per course. Patients with a positive LP receive methotrexate IT or intraventricularly OR cytarabine IT or intraventricularly OR methotrexate IT or intraventricularly, cytarabine IT or intraventricularly, and therapeutic hydrocortisone IT or intraventricularly.
  MAINTENANCE:
  Patients not treated with consolidative SCT, receive ixazomib citrate PO BID on days 1, 8, and 15. Treatment repeats every 28 days for up to one year in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Cytarabine: Given IT or intraventricularly
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ixazomib Citrate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IT or intraventricularly
  Prednisone: Given PO
  Rituximab: Given IV
  Therapeutic Hydrocortisone: Given IT or intraventricularly
  Vincristine Sulfate: Given IV
Arm/Group | Treatment (Combination Chemotherapy, Rituximab, Ixazomib)
Number analyzed (Participants) | 5
mg | 3

2. Primary Outcome: 12-month PFS (Progression Free Survival) of Treatment With Ixazomib in Combination With DA-EPOCH-R (Phase II)
Description: 12-month PFS will be defined as the percentage of patients alive and progression free 12 months from start of therapy. Patients lost to follow up will be censored from last point of contact. PFS was calculated using a Kplan-meier estimation with the probability of patients being progression free at 12 months, presented as the percentage based on this probability.
Time Frame: Up to 12 months from initiation of treatment
Population: Only patients included in the phase II dose are included in this endpoint per protocol.
Measure: Number (95% Confidence Interval); unit: probability (%) of patients alive
Arm/Group | Treatment (Combination Chemotherapy, Rituximab, Ixazomib)
Number analyzed (Participants) | 36
probability (%) of patients alive | 75.84 [62.50 to 92.03]

3. Secondary Outcome: Toxicity of Treatment With Ixazomib in Combination With DA-EPOCH-R
Description: Adverse events will be assessed using CTCAE v 4.03.
  In general grading will be as follows:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities.
  Moderate (grade 2): the event causes discomfort that affects normal daily activities.
  Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Life-threatening (grade 4): the patient was at risk of death at the time of the event.
  Fatal (grade 5): the event caused death.
Time Frame: Assessed at the beginning each cycle with up to 6 cycles of induction treatment and up to 13 cycles of maintenance treatment (1 cycle =21 days) and at approximately 21 days after the last treatment.
Reporting Status: Not Posted, anticipated posting 2023-12

4. Secondary Outcome: Overall Survival (OS)
Description: OS will be defined as freedom from death by any cause and measured from time of treatment initiation and completion of follow up or death from any cause.
Time Frame: Up to approximately 30 months
Reporting Status: Not Posted, anticipated posting 2023-12

5. Secondary Outcome: Response Rate
Description: Anti-tumor activity will be defined as the detection of SD (Stable Disease), Partial Response (PR), or CR (Complete Remission) by CT or PET/CT scan, and/or resolution of marrow-only involvement. CR and PR will each be assessed according to the Revised Response Criteria for Malignant Lymphoma. Assessments will be performed after cycles 2 and 6, then at the discretion of the investigator.
  In general:
  CR-Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms PR-At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. No increase should be observed in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by ≥50% in their SPD or, for single nodules, in the greatest transverse diameter. No new sites of disease should be observed.
  SD-fails to attain the criteria needed for a CR or PR, but does not fulfill those for progressive disease
Time Frame: After 2 cycles, then after 6 cycles and then at the discretion of the investigator for up to 13 maintenance cycles (1 cycle = 21 days)
Reporting Status: Not Posted, anticipated posting 2023-12

6. Secondary Outcome: Assess the Predictive Value of FDG-PET/CT Scans on PFS
Description: Patients will be categorized as either FDG-PET (+) or (-) at interim and end-of treatment imaging.
Time Frame: Up to 1 year after treatment stopped
Reporting Status: Not Posted, anticipated posting 2023-12

7. Other Pre Specified Outcome: Determine the Impact of Cell of Origin (COO) Upon Response Rate, PFS, and OS
Description: Impact of COO defined as germinal center B-cell (GCB) and non-GCB via the Hans algorithm upon response rate, PFS, and OS (applicable only to patients with DLBCL).
Time Frame: Up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Consolidation SCT (Stem Cell Transplant)
Description: Feasibility and outcomes of consolidation SCT will be assessed. Patients will be grouped by whether consolidative SCT was performed in first remission, with PFS compared across groups (SCT vs. non-SCT).
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the beginning of each cycle for up to 6 induction cycles and up to 13 maintenance cycles (1 cycle = 21 days) and 21 days after the last study treatment
Description: Secondary endpoints are written to have phase I & II patient data combined in analysis. Due to the way that adverse event data collected was analysed (i.e. phase I/II data was analysed combined regardless of dose) all patients data here is shown as one cohort regardless of initial dose of ixazomib given. This is due to the way the protocol was written and that only 2 patients out of 38 received a different initial starting dose (and the starting dose for all in maintenance was 4 mg).
Arm/Group | Treatment (Combination Chemotherapy, Rituximab, Ixazomib)
All-Cause Mortality (participants affected / at risk) | 6/38
Serious Adverse Events (participants affected / at risk) | 20/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy, Rituximab, Ixazomib) (N=38)
Cholecystitis (Infections and infestations) | 1 (1) — patient experienced influenza B infection at the same time as the SAE
Lung infection (Infections and infestations) | 1 (1) — Patient also experienced anemia, febrile neutropenia, weakness and dehydration at the same time of the SAE
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 (8)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) — Patient also with febrile neutropenia at the same time as this event.
duodenitis (Infections and infestations) | 1 (1)
Spinal fracture (lumbar) (Injury, poisoning and procedural complications) | 1 (1) — Patient also with back pain at the time of this event
Sepsis (Infections and infestations) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
parainfluenza 3 (Infections and infestations) | 1 (1) — Patient also with pneumonia and lung infection at the time of this event
Thromboembolic event - pulmonary embolism (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also with lung infection and hypoxia at the time of the event
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Patient also with Muscle weakness, lower limbs, bilateral at the time of the event
Cardiac Arrest (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) — Patient also with Urinary tract infection at the same time as the event
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Patient also with Febrile neutropenia at the same time as the event
Small intestine and colonic perforation (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) — Patietn also with colonic obstruction an constipation at the time of the event
gastric adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient also with febrile neutropenia at the time of the event
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Patient also with back pain at the time of the event
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Combination Chemotherapy, Rituximab, Ixazomib) (N=38)
Anemia (Blood and lymphatic system disorders) | 38
Lymphocyte count decreased (Investigations) | 38
Platelet count decreased (Investigations) | 38
Hypoalbuminemia (Metabolism and nutrition disorders) | 37
Fatigue (General disorders) | 35
Hypertension (Vascular disorders) | 34
Hypocalcemia (Metabolism and nutrition disorders) | 34
White blood cell decreased (Investigations) | 34
Hypokalemia (Metabolism and nutrition disorders) | 33
Neutrophil count decreased (Investigations) | 33
Constipation (Gastrointestinal disorders) | 32
Peripheral sensory neuropathy (Nervous system disorders) | 30
Nausea (Gastrointestinal disorders) | 29
Alkaline phosphatase increased (Investigations) | 24
Hyperglycemia (Metabolism and nutrition disorders) | 24
Hypophosphatemia (Metabolism and nutrition disorders) | 24
Alanine aminotransferase increased (Investigations) | 22
Mucositis oral (Gastrointestinal disorders) | 22
Weight loss (Investigations) | 22
Aspartate aminotransferase increased (Investigations) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Edema limbs (General disorders) | 20
Headache (Nervous system disorders) | 20
Hyponatremia (Metabolism and nutrition disorders) | 20
Diarrhea (Gastrointestinal disorders) | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Anxiety (Psychiatric disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 16
Vomiting (Gastrointestinal disorders) | 16
Dysgeusia (Nervous system disorders) | 15
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15
Pain (General disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 14
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 13
Investigations - Other, specify (Investigations) | 13
Creatinine increased (Investigations) | 12
Depression (Psychiatric disorders) | 12
Sinus tachycardia (Cardiac disorders) | 12
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Chills (General disorders) | 10
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10
Hypernatremia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Cardiac disorders - Other, specify (Cardiac disorders) | 9
Fever (General disorders) | 9
General disorders and administration site conditions - Other, specify (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 9
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9
Blood bilirubin increased (Investigations) | 8
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 8
Localized edema (General disorders) | 8
Paresthesia (Nervous system disorders) | 8
Urinary frequency (Renal and urinary disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 7
Bruising (Injury, poisoning and procedural complications) | 7
Hemorrhoids (Gastrointestinal disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7
Infections and infestations - Other, specify (Infections and infestations) | 7
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 7
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 7
Dry mouth (Gastrointestinal disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 6
Hyperuricemia (Metabolism and nutrition disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 5
Blurred vision (Eye disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Eye disorders - Other, specify (Eye disorders) | 5
Infusion related reaction (General disorders) | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 5
Thromboembolic event (Vascular disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Hypotension (Vascular disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Non-cardiac chest pain (General disorders) | 4
Obesity (Metabolism and nutrition disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 4
Tremor (Nervous system disorders) | 4
Urinary tract infection (Infections and infestations) | 4
Weight gain (Investigations) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Bloating (Gastrointestinal disorders) | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Cataract (Eye disorders) | 3
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Hot flashes (Vascular disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
INR increased (Investigations) | 3
Lethargy (Nervous system disorders) | 3
Lymph node pain (Blood and lymphatic system disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Nail loss (Skin and subcutaneous tissue disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Sepsis (Infections and infestations) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 3
Upper respiratory infection (Infections and infestations) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Cholesterol high (Investigations) | 2
Confusion (Psychiatric disorders) | 2
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Immune system disorders - Other, specify (Immune system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 2
Lung infection (Infections and infestations) | 2
Malaise (General disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Palpitations (Cardiac disorders) | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Retinal detachment (Eye disorders) | 2
Sinusitis (Infections and infestations) | 2
Toothache (Gastrointestinal disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Watering eyes (Eye disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Aphonia (Nervous system disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Delirium (Psychiatric disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Esophageal infection (Infections and infestations) | 1
Eye pain (Eye disorders) | 1
Facial pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infusion site extravasation (General disorders) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lymphedema (Vascular disorders) | 1
Lymphocyte count increased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 1
Presyncope (Nervous system disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus pain (Nervous system disorders) | 1
Skin infection (Infections and infestations) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Urine output decreased (Investigations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Vitreous hemorrhage (Eye disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Wound infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study closed accrual prior to the planned sample size being enrolled and treated on the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02481310/Prot_SAP_000.pdf